CLINICAL TRIAL: NCT00374218
Title: Effect of Replacing HFCS With Sucromalt on Glucose Tolerance, Blood Lipids and Inflammatory Markers in Subjects With Raised Waist Circumference
Brief Title: Effect of Replacing HFCS With Sucromalt in Subjects With Raised Waist Circumference
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UTREB17491
Record Dates: First submitted 2006-09-08; First posted 2006-09-11 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Abdominal Obesity
Keywords: Carbohydrate; Glycemic index; Randomized; Double-blind; Glucose; Insulin; C-reactive protein
MeSH Terms: conditions — Obesity, Abdominal; Insulin Resistance | interventions — High Fructose Corn Syrup; sucromalt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: High Fructose Corn Syrup
Drug: Sucromalt

SUMMARY:
Weight gain is linked to a high consumption of soft-drinks and other beverages sweetened with high fructose corn syrup. Being overweight increases risk for diabetes and heart disease. These problems may be due to high blood glucose and insulin responses caused by high fructose corn syrup. Sucromalt is a sweetener which contains the same amount of carbohydrate at high fructose corn syrup, but causes lower glucose and insulin responses. The purpose of this study is to see if consuming soft-drinks and other foods sweetened with sucromalt instead of high fructose corn syrup will result in lower levels of blood glucose, insulin, cholesterol and other markers of risk. We are including in this study people who are overweight and normally consume soft-drinks because they are the ones most likely to benefit from this change.

DETAILED DESCRIPTION:
Diets with a high glycemic load (GL) are associated with increased risk of diabetes and cardiovascular disease, possibly because of their association with the metabolic syndrome, dyslipidemia and increased markers of chronic inflammation. Since GL is the product of glycemic index (GI) times the amount of carbohydrate in the diet, GL can be reduced either by reducing GI or by reducing carbohydrate intake, and the effect of these maneuvers on health biomarkers may not necessarily be the same.

A high consumption of sugars in regular soft drinks has been associated with increased weight gain in adolescents, and, in adults, replacing starch with sucrose in the diet has been shown to result in weight gain and an increase in blood pressure and certain inflammatory markers. However, in the latter studies, the effects of sucrose in sucrose-sweetened beverages and foods were compared to those of aspartame-sweetened beverages and foods. Since aspartame contains no energy, the sucrose and control diets differed not only in sucrose, but also in energy, fat and protein; with more energy and less fat and protein as a % of energy on the sucrose than the control diet. This results in a problem in interpretation of the results because it is not possible to know what dietary change was responsible for the changes in biomarkers - indeed some changes due to increased sucrose intake may have been offset by opposite changes in, for example, saturated fat intake.

Another approach to studying the effect of reducing the GL of the diet is to reduce the GI of the diet without changing the amounts of energy, carbohydrate, fat or protein. Such an approach may be more scientifically desirable because it is possible to study the effect of changing only one dietary variable. Recently, the development of sucromalt allows the replacement of high fructose corn syrup (HFCS) in foods and beverages with a nutritive carbohydrate sweetener that has a reduced GI. Sucromalt is an enzymatically modified carbohydrate which we have shown elicits lower glucose and insulin responses than HFCS without apparent malabsorption. Therefore, the purpose of this study is to conduct a pilot study to see if exchanging HFCS with sucromalt has any effect on glucose tolerance and fasting blood lipids and inflammatory biomarkers in subjects with a high waist circumference.

ELIGIBILITY:
Inclusion Criteria:

* males or non-pregnant and non-lactating females
* aged 20-50
* normally drink at least 2 cans (680ml) regular soft-drinks or sugar sweetened drinks per day
* high waist circumference (≥102cm (40in) in men or ≥88cm (34.5in) in women)

Exclusion Criteria:

* Body mass index >35.0kg/m²
* Subjects whose weight is not stable (varied by >5% of current weight over the past 6 months).
* Subject who regularly undertake >30min vigorous physical activity per week.
* Diabetes based on current treatment with insulin or an oral hypoglycemic agent or fasting glucose ≥7.0mmol/L on screening
* Fasting triglycerides ≥10.0mmol/L
* Severe liver dysfunction (transaminase >180% of upper limit of normal)
* Severe renal impairment (serum creatinine >140% of upper limit of normal)
* Any major medical or surgical event within 6 months
* History of inflammatory bowel disease, malabsorption, or other disorder or drug use affecting gastrointestinal motility or the absorption of nutrients
* Use of drugs which affect glucose or lipids except: stable doses (3 months) of statins, fibrates, beta-blockers, diuretics.
* Substance abuse
* Simultaneous participation in another clinical trial
* Any other condition which, in the opinion of Dr. Wolever, might make the subject's participating harmful to him(her)self or others or affect the results
* Inability to understand spoken and written English
* Unwilling or unable to consume the test foods (drinks and nutrition bars) and/or to undergo the test procedures
* Unwilling or unable to give informed consent and/or sign the consent form

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2006-09; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Fasting and 2h glucose after 75g oral glucose tolerance test | 4 weeks

SECONDARY OUTCOMES:
Fasting and 2h insulin after 75g oral glucose | 4 weeks
Gut hormone responses (eg. GLP-1) after 75g oral glucose | 4 weeks
Postprandial glucose and insulin elicited by control and test foods/drinks | Baseline
Fasting blood lipids (total, HDL and LDL cholesterol and triglycerides) | Baseline and 4 weeks
Fasting C-reactive protein | Baseline and 4 weeks
Fasting apolipoproteins A1 and B100 | Baseline and 4 weeks
Body weight | Weekly for 4 weeks
Waist circumference | 4 weeks
Blood pressure | 4 weeks
Symptoms | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Glycemic Index Laboratories, Toronto, Ontario, Canada